CLINICAL TRIAL: NCT01452555
Title: Video-Based Delivery of HIV Test Information for Spanish-Speaking Latinos
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21NR011997 (NIH)
Record Dates: First submitted 2011-10-06; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-08

CONDITIONS: HIV; AIDS
Keywords: HIV; HIV Prevention; HIV testing; HIV Rapid Test
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- In Person Counseling (Active Comparator): Participants will receive an in person HIV and HIV testing counseling session
  Interventions: Behavioral: Video or In-Person Presentation
- Video Presentation (Experimental): Participants will watch an HIV and HIV testing video
  Interventions: Behavioral: Video or In-Person Presentation

INTERVENTIONS:
Behavioral: Video or In-Person Presentation — Participants will be randomly assigned to an in person counseling session or will watch a HIV and HIV testing video

SUMMARY:
The purpose of the study is to determine if a Spanish-language HIV and HIV test information video is as effective in delivering basic information regarding HIV and HIV tests to primarily Spanish-speaking HIV test recipients as an in-person presentation with an HIV test counselor.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* Self-identify as Latino
* Able to give informed consent
* Spanish speaking

Exclusion Criteria:

* Intoxicated
* Being treated for acute psychiatric illness
* Mental incapacitation
* Significant visual or hearing impairment
* Prisoner or under home confinement
* Participating in HIV vaccine trial
* Critically ill

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08

PRIMARY OUTCOMES:
Effectiveness of an educational video regarding HIV and HIV testing for Spanish speaking Latinos
  Participants in both arms will complete an HIV knowledge questionnaire after recieving an in-person presentation or watching the video to compare the effectiveness of an HIV educational video for Spanish speaking Latinos regarding HIV and HIV tests.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Roland Merchant, MD, MPH, ScD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Merchant RC, Clark MA, Santelices CA, Liu T, Cortes DE. Efficacy of an HIV/AIDS and HIV testing video for Spanish-speaking Latinos in healthcare and non-healthcare settings. AIDS Behav. 2015 Mar;19(3):523-35. doi: 10.1007/s10461-014-0889-6. PMID 25179540